CLINICAL TRIAL: NCT04874870
Title: Clinical Effectiveness of Splinting After Collagenase Clostridium Histolyticum Injection for Dupuytren Contracture
Brief Title: Effectiveness of Splinting After Collagenase Injection
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Foundation for Orthopaedic Research and Education (Other)
Collaborators: Endo, Inc. (Unknown)
Responsible Party: Principal Investigator, Jason Nydick DO, Jason Nydick DO, Foundation for Orthopaedic Research and Education
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FORE- CHI 2021
Record Dates: First submitted 2021-04-23; First posted 2021-05-06 (Actual); Last update posted 2025-02-26 (Actual); Status verified 2025-02

CONDITIONS: Dupuytren Contracture; Dupuytren's Disease
MeSH Terms: conditions — Dupuytren Contracture | interventions — Microbial Collagenase

STUDY DESIGN:
Intervention Model Description: Randomized, Controlled
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- No Splint Group (Active Comparator): This group will receive Xiaflex injection only
  Interventions: Drug: Collagenase Clostridium Histolyticum 0.9 MG [Xiaflex]
- Splint Group (Active Comparator): This group will receive Xiaflex injection and hand-based custom orthosis to maintain finger extension
  Interventions: Combination Product: Xiaflex + Hand-Based Custom Orthosis

INTERVENTIONS:
Drug: Collagenase Clostridium Histolyticum 0.9 MG [Xiaflex] — 1 injection of 0.58mg will be injected into applicable cord.
  Other Names: Xiaflex
  Arms: No Splint Group
Combination Product: Xiaflex + Hand-Based Custom Orthosis — 1 injection of 0.58mg will be injected into applicable cord followed by use of hand-based custom orthosis to maintain finger extension
  Arms: Splint Group

SUMMARY:
Dupuytren disease is a fibroproliferative condition of the palmar and digital fascia. A collagen containing cord forms which can lead to fixed flexion contracture of one or more fingers. While there is no cure, many treatment options are available to manage symptoms. One of these options is injectable collagenase clostridium histolyticum (CCH). CCH is a combination of two highly selective microbial collagenases that can disrupt collagen types I and III usually found in cords. Current standard of care after receiving a CCH injection is daily hand exercises and use of a static night brace for four months. However, there is limited evidence that use of a night splint after CCH injection has any benefit post-treatment. The goal of our randomized, controlled trial, is to determine the clinical effectiveness of splinting after CCH injection. Study subjects will be adults 18 years of age or older with Dupuytren disease and contracture of one or more digits. Treatment includes collagenase clostridium histolyticum injection for Dupuytren flexion contraction, with randomization to static night splint or no splint.

DETAILED DESCRIPTION:
Patients with Dupuytren disease that meet inclusion criteria will be consented to participate. All patients will be randomized to splint or no splint group prior to treatment. Baseline data will be collected prior to treatment and will include demographics, measurement of joint flexion contracture(s) with a standard finger goniometer, and QuickDASH scores. All patients that participate will receive 1 injection of 0.58 mg of CCH into cord. After 24-48 hours, if needed, patient will return to clinic for extension manipulation of treated finger(s) to help facilitate rupture of cord. Following injection and/or manipulation, all patients will be instructed to perform a series of finger exercises daily that they will receive from a hand therapist. In addition, patients assigned to the splint group will be fitted for a static night splint that they will be instructed to wear nightly for 4 months. Splint compliance will be recorded by a survey at each follow up visit. Patients will return to clinic for routine follow up care at 1 month and 4 months during which their degree of contracture(s) and outcomes will be measured and recorded. The primary outcome measures of this study are improvement in active extension deficit of each joint and total active extension of each digit, in degrees. The secondary outcome measures are QuickDASH scores and patient satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Contracture of 1 or more digits caused by palpable cord
* PIP joint flexion contracture of 20 degrees or more or;
* MCP joint flexion contracture of 20 degrees or more

Exclusion Criteria:

* Age less than 18 years
* Prior CCH injection for contracture less than 1 year before start of study
* Prior surgical intervention for contracture less than 1 year before start of study

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2021-07-12 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2023-12-01 (Actual)

PRIMARY OUTCOMES:
Improvement in active extension deficit of MCP joint, in degrees, if applicable | Baseline, 1 month, and 4 months
  Clinical measurement of MCP joint extension with goniometer, in degrees, of treated finger
Improvement in active extension deficit of PIP joint, in degrees, if applicable | Baseline, 1 month, and 4 months
  Clinical measurement of PIP joint extension with goniometer, in degrees, of treated finger
Improvement in total active extension of each digit, in degrees | Baseline, 1 month, and 4 months
  Sum of MCP and PIP joint extension, in degrees, of treated finger

SECONDARY OUTCOMES:
Compliance of Splint wearing (Splint group only) | 1 month and 4 months
  By compliance survey composed of 4 items
  Items 1 and 2 scored from 1-5; 1 - not at all, 2 - slightly, 3- moderately, 4- very, 5- extremely
  How comfortable was your splint?
  Was the splint easy to use?
  Items 3 and 4 scored from 1-5; 1 - not at all, 2 - occasionally, 3- half of the time, 4 - most of the time, 5 - all of the time
  Did you wear your splint every night?
  Did you have any issues with your splint?
Functional Outcomes | Baseline, 1 month, and 4 months
  Quick Disabilities of the Arm, Shoulder, and Hand (QuickDASH) questionnaire score will be used to measure clinical outcomes. The QuickDASH is scored in two components: the disability/symptom section (11 items, scored 1-5) and the optional high performance sport/music or work modules (four items, scored 1-5). From the item scores, scale scores are calculated, ranging from 0 (no disability) to 100 (most severe disability).
Patient Satisfaction | 1 month and 4 months
  By satisfaction scale composed of 3 items (each of them scored from 1-5; 1 - not at all, 2 - slightly, 3- moderately, 4- very, 5- extremely)
  How satisfied are you with the progress of your hand?
  How satisfied are you with your treatment?
  Has your quality of life improved?

CONTACTS AND LOCATIONS:
Overall Officials: Jason Nydick, DO, Principal Investigator — Florida Orthopaedic Institute
Locations (1):
- Florida Orthopaedic Institute, Tampa, Florida, United States

IPD SHARING:
Plan to Share IPD: No
Pending results- the plan would be to submit a poster for presentation and a manuscript for publication.

REFERENCES:
- [Background] Rayan GM. Dupuytren disease: Anatomy, pathology, presentation, and treatment. J Bone Joint Surg Am. 2007 Jan;89(1):189-98. doi: 10.2106/00004623-200701000-00026. No abstract available. PMID 17256226
- [Background] Hurst LC, Badalamente MA, Hentz VR, Hotchkiss RN, Kaplan FT, Meals RA, Smith TM, Rodzvilla J; CORD I Study Group. Injectable collagenase clostridium histolyticum for Dupuytren's contracture. N Engl J Med. 2009 Sep 3;361(10):968-79. doi: 10.1056/NEJMoa0810866. PMID 19726771
- [Background] Bowers NL, Merrell GA, Foster T, Kaplan FTD. Does Use of a Night Extension Orthosis Improve Outcomes in Patients With Dupuytren Contracture Treated With Injectable Collagenase? J Hand Surg Glob Online. 2021 Jun 26;3(5):272-277. doi: 10.1016/j.jhsg.2021.05.001. eCollection 2021 Sep. PMID 35415567